CLINICAL TRIAL: NCT06111313
Title: A Phase 2 Risk Adapted Parallel Randomized Trial of MRI-Guided Lattice Stereotactic Focal Radiotherapy of the Prostate With or Without Ultra-Short Term Androgen Deprivation Therapy-The Miami UAdapt Trial
Brief Title: The University of Miami Adapt (UAdapt) Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Principal Investigator, Benjamin Spieler, Assistant Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20230097
Record Dates: First submitted 2023-10-26; First posted 2023-11-01 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — relugolix

STUDY DESIGN:
Intervention Model Description: The Miami UAdapt Trial is a non-comparative phase II study that includes two parallel randomized cohorts that will prospectively assign men radiotherapy (RT) treatment. Patients with relatively favorable risk prostate cancer (PCa) will be eligible for focal therapy LEAD (FTLEAD) RT (n=40), and randomized to receive Lattice Extreme Ablative Dose (LEAD) single high dose RT (SDRT, 12-16 Gy) vs. the same overall plan with the addition of ultrashort-term ADT (uSTADT, 1 month duration) concurrent with SDRT. Higher risk patients are assigned to the HypoLEAD cohort (n=90) and randomized 1:1 to receive Lattice Extreme Ablative Dose (LEAD) single high dose RT (SDRT, 16-20 Gy) followed by moderately hypofractionated (HypoFx) RT for 25 additional fractions vs. the same overall plan with the addition of ultrashort-term ADT (uSTADT, 1 month duration) concurrent with SDRT. In HypoLEAD additional ADT will be assigned at physician discretion per standard of care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Focal Therapy lattice extreme ablative dose (FTLEAD), RT Only, Arm A (Experimental): Participants in this group will receive the FTLEAD treatment only and will be followed for up to 5.5 years.
  Interventions: Radiation: FTLEAD
- Focal Therapy lattice extreme ablative dose (FTLEAD), uSTADT, Arm B (Experimental): Participants in this group will receive the FTLEAD treatment and ultra short-term androgen deprivation therapy (ADT) and will be followed for up to 5.5 years.
  Interventions: Radiation: FTLEAD; Drug: Ultra-Short-Term Androgen Deprivation Therapy with Relugolix
- Lattice extreme ablative dose followed by hypofractionated RT (HypoLEAD), Arm C (Experimental): Participants in this group will receive LEAD RT followed by moderately hypofractionated RT (HypoLEAD) and standard of care androgen deprivation therapy and will be followed for 5.5-8 years.
  Interventions: Radiation: FTLEAD; Radiation: HypoLEAD; Drug: ADT Standard of Care
- Lattice extreme ablative dose followed by hypofractionated RT (HypoLEAD), uSTADT, Arm D (Experimental): Participants in this group will receive LEAD RT with ultra short-term ADT followed by moderately hypofractionated RT (HypoLEAD) and standard of care ADT and will be followed for 5.5-8 years.
  Interventions: Radiation: FTLEAD; Drug: Ultra-Short-Term Androgen Deprivation Therapy with Relugolix; Radiation: HypoLEAD; Drug: ADT Standard of Care

INTERVENTIONS:
Radiation: FTLEAD — In focal therapy lattice extreme ablative (FTLEAD) RT, the multiparametric-MRI (mpMRI) defined gross tumor volume (GTV) will receive 16-20 Gy in a single fraction of RT to the targeted area which is the tumor within the prostate, with or without uSTADT.
Drug: Ultra-Short-Term Androgen Deprivation Therapy with Relugolix — Ultra-Short-Term Androgen Deprivation Therapy (uSTADT) is hormone therapy that includes Relugolix. Patients will receive a loading dose of uSTADT for a total duration 4 weeks (28 days), with oral LHRH antagonist relugolix administered daily starting 2 weeks prior to LEAD RT and continuing until 2 weeks afterwards as per Study Calendar. Patients randomized to uSTADT will receive a loading dose of 360 mg of oral relugolix on Day 14 followed by 120 mg of oral relugolix daily from Day 13 to Day 14. Patients will be instructed to take relugolix orally once daily at approximately the same time each day. Patients may take relugolix with or without food and should swallow tablets whole and not crush or chew tablets.
  Arms: Focal Therapy lattice extreme ablative dose (FTLEAD), uSTADT, Arm B; Lattice extreme ablative dose followed by hypofractionated RT (HypoLEAD), uSTADT, Arm D
Radiation: HypoLEAD — In Hypofractionated LEAD (HypoLEAD), the multiparametric-MRI (mpMRI) defined GTV will receive 12-16 Gy in a single fraction on the first day of treatment, with or without uSTADT. Four weeks after LEAD RT, patients will begin whole prostate moderately hypoLEAD (67.5 Gy in 25 fractions) with pelvic nodal irradiation and further ADT at the discretion of the treating physician.
  Arms: Lattice extreme ablative dose followed by hypofractionated RT (HypoLEAD), Arm C; Lattice extreme ablative dose followed by hypofractionated RT (HypoLEAD), uSTADT, Arm D
Drug: ADT Standard of Care — Participants will receive ADT as per standard of care (SOC).
  Arms: Lattice extreme ablative dose followed by hypofractionated RT (HypoLEAD), Arm C; Lattice extreme ablative dose followed by hypofractionated RT (HypoLEAD), uSTADT, Arm D

SUMMARY:
The Miami UAdapt Trial is a non-comparative, risk adapted, parallel, randomized, phase 2 study for patients with favorable-intermediate to very high risk non-metastatic prostate cancer with the primary objective of assessing the efficacy and modulation of response of Lattice Extreme Ablative Dose (LEAD) RT with and without androgen deprivation therapy (ADT) at a multidimensional level.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy confirmed adenocarcinoma of the prostate (including intraductal adenocarcinoma, excluding small cell carcinoma).
2. T1-T3 disease based on digital rectal exam (DRE), informed by mpMRI. Prostate MRI may aid in the staging evaluation by verifying organ-confined status6,7. The ability to distinguish between organ-confined tumors (≤T2c) and those that extend beyond the prostate (≥T3a) is an important component of treatment decision making.
3. Patients with T3 disease based on DRE, mpMRI, Gleason 8-10, or a PSA of >15 ng/mL, should undergo a negative metastatic workup prior to signing of consent. A questionable bone scan is acceptable if additional imaging studies; eg, plain x-rays, CT, MRI, prostate specific membrane antigen (PSMA) positron emission tomography (PET)/CT do not confirm for metastasis.
4. No evidence of metastasis by clinical criteria or available radiographic tests (N0M0 by clinical or imaging criteria).
5. Gleason score 6-10.
6. Prostate specific antigen (PSA) ≤100 ng/mL within (≤) 3 months of signing of consent. If PSA was above 100 ng/mL and drops to ≤100 ng/mL with antibiotics, this is acceptable for enrollment.
7. Suspicious peripheral zone or central gland lesion(s) on mpMRI.

   1. Peripheral zone: Distinct lesion on dynamic contrast enhanced (DCE)-MRI with early enhancement and later washout (Note: contrast not required for enrollment), and/or distinct lesion on the apparent diffusion coefficient (ADC) map (Value <1000).
   2. Central gland: A suspicious central gland lesion on mpMRI must have a distinct lesion on the ADC map (Value <1000).
8. No previous pelvic radiotherapy.
9. No previous history of radical/total prostatectomy (suprapubic prostatectomy is acceptable).
10. No concurrent, active malignancy, other than nonmetastatic skin cancer or early-stage chronic lymphocytic leukemia (well-differentiated small cell lymphocytic lymphoma). If a prior malignancy is in remission for ≥5 years, then the patient is eligible.
11. Ability to understand and the willingness to sign a written informed consent document.
12. Zubrod performance status ≤2. Karnofsky or Eastern Cooperative Oncology Group (ECOG) performance status may be used to estimate Zubrod.
13. Age ≥35 and ≤85 years at signing of consent.
14. Serum testosterone is within 40% of normal assay limits (eg, x=0.4*lower assay limit and x=0.4*upper assay limit + upper assay limit), taken within (≤) 3 months of signing of consent.
15. For patients in HypoLEAD cohort, post-LEAD RT androgen deprivation therapy, including use of secondary agents (eg, abiraterone), is at the discretion of the treating physician but must be declared as none, short-term or long-term prior to enrollment. Note that this ADT regimen differs from the uSTADT regimen. If antiandrogen therapy (eg, bicalutamide) or ADT (LHRH agonist or antagonist injection) is planned, the following restrictions apply:

    1. Anti-androgen therapy and ADT must be started after 3-week post-LEAD RT gradient biopsy.
    2. Anti-androgen therapy and ADT are recommended to be started prior to or concurrent with start of moderately hypofractionated RT course and must be started before the end of the hypofractionated RT course.
    3. The total length planned must be ≤ 30 months.
16. Patient unable to receive iodine or gadolinium contrast due to allergy or poor renal function are still eligible for enrollment.

Exclusion Criteria:

1. Prior pelvic radiotherapy.
2. Prior androgen ablation therapy.
3. Prior or planned radical prostate surgery.
4. Clinical, radiographic, or pathologic evidence of nodal or distant metastatic disease with the following specifications: PSMA-PET or Fluciclovine PET: Patients with subclinical (<1.5 cm) pelvic lymph nodes that are suspicious on such PET scans will be ineligible for FTLEAD, however will still be eligible for HypoLEAD. In the latter case the treating physician may boost such nodes to a higher dose.
5. Concurrent, active malignancy, other than nonmetastatic skin cancer or early-stage chronic lymphocytic leukemia (well-differentiated small cell lymphocytic lymphoma). If a prior malignancy is in remission for > 5 years, then the patient is eligible.
6. Zubrod status >2.
7. Pretreatment PSA >100 ng/ml or Gleason score <6. If PSA was above 100 ng/mL and drops to ≤100 ng/mL with antibiotics, this is acceptable for enrollment.
8. Thyroxine (T4) disease.
9. Patients with impaired decision-making capacity who lack the ability to understand and voluntarily sign a written informed consent document.
10. Patients unable to tolerate diagnostic MRI acquisition. Note: inability to tolerate contrast agents is not exclusionary.

Ages: 35 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2033-11-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of Patients with Biochemical Disease Failure (FFBN9mo) | Up to 14 Months
  Biochemical Disease Failure will be determined by the proportion of patients with biochemical disease failure.
Proportion of Patients with Clinical Disease Failure | Up to 14 Months
  Clinical Disease Failure will be determined by the proportion of patients with clinical disease failure. Clinical disease failure will include the proportion of patients with biopsy finding of treatment failure.

SECONDARY OUTCOMES:
Proportion of Patients with Biochemical Disease Failure (Phoenix definition) | Up to 2.5 years
  Biochemical Disease Failure will be determined by the proportion of patients with biochemical disease failure.
Proportion of Patients with Clinical Disease Failure | Up to 2.5 years
  Clinical Disease Failure will be determined by the proportion of patients with clinical disease failure. Clinical disease failure will include the proportion of patients with biopsy finding of treatment failure.
Proportion of Patients with Pathology-determined complete response (PathCR) | Up to 2.0-2.5 years after all treatment
  Pathology-determined complete response (PathCR) is defined as proportion of patients with negative prostate biopsy findings on both template plus image-guided habitat biopsy.
Proportion of Patients with Pathology-determined complete response (PathCR) | Up to 2.5 year
  Pathology-determined complete response (PathCR) is defined as proportion of patients with negative prostate biopsy findings on both template plus image-guided habitat biopsy.
Incidence of Failure rate (FR) | Up to 2.5 years
  Failure rate is defined as the cumulative incidence of biopsy finding of treatment failure (BxTF), biochemical failure (BF), or clinical failure (CF), or combined (BxTF plus BF plus CF), where combined failure refers to documented evidence of BxTF, BF, and CF occurring within 6 months of each other with the earlier date used, or death related to prostate cancer without prior evidence of failure, whichever is earlier, from study enrollment allowing for competing risk as needed.
Number of Treatment Related Acute toxicity | Up to 3 months
  Acute toxicity is defined as grade 2+ and grade 3+ treatment-related acute genitourinary (GU)/gastrointestinal (GI) toxicity occurring during treatment and within 3 months of completing treatment. The severity of the reactions to treatment will be scored according to the criteria outline in CTCAE version 5.0.
Number of Treatment Related Late toxicity | Up to 8 Years
  Late toxicity is defined as grade 2+ and grade 3+ treatment-related GU/GI toxicity occurring more than 3 months after completing study treatment. The severity of the reactions to treatment will be scored according to the criteria outline in CTCAE version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Spieler, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No